CLINICAL TRIAL: NCT01023373
Title: Phase 4 Study of Medical Therapy Versus Medical Therapy Plus Renal Artery Stenting in Preventing the Progression of Renal Failure in Atherosclerotic Renovascular Disease
Brief Title: Revascularization of Renal Artery Stenosis Versus Medical Therapy for the Treatment of Ischemic Nephropathy
Acronym: NITER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Roberto Scarpioni, MD, Divisione Nefrologia e Dialisi, da Saliceto Hospital, AUSL Piacenza, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 388-2002
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Atherosclerosis; Chronic Kidney Disease; Hypertension, Renovascular; Ischemic Nephropathy; Renal Artery Stenosis
Keywords: Angioplasty; Atherosclerotic reno vascular disease (ARVD); Cardio- and cerebro- vascular comorbidity; End stage renal disease (ERSD); kidney diseases; High blood pressure; Hypertension; Ischemic nephropathy; Percutaneous transluminal renal artery stenting (PTRS); Randomized controlled trials; Renal artery stenosis (RAS); Renal insufficiency; Vascular diseases
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic; Hypertension, Renovascular; Renal Artery Obstruction; Kidney Failure, Chronic; Kidney Diseases; Hypertension; Renal Insufficiency; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B:PTRS (Experimental): B: the same medical therapy, as previously described in group A, associated with PTRS
  Interventions: Procedure: PTRS; Device: renal artery stent
- A:medical therapy (Active Comparator): hypotensive drugs, statins and antiplatelet therapy
  Interventions: Drug: Medical treatment; Device: renal artery stent

INTERVENTIONS:
Drug: Medical treatment — hypotensive drugs, statins and anti-platelets
  Arms: A:medical therapy
Procedure: PTRS — Percutaneous transluminal renal artery stenting. The same medical therapy, as in group A, plus PTRS
  Arms: B:PTRS
Device: renal artery stent — Non-drug intervention, percutaneous transluminal renal artery stent angioplasty
  Arms: B:PTRS
Device: renal artery stent — Adding the renal artery stenting (in group B) to the optimal medical therapy (as in group A) that includes hypotensive drugs, statins and antiplatelet therapy

SUMMARY:
The aim of the study is to value, in patients with chronic kidney disease and hypertension, whether medical therapy plus interventional renal artery revascularization is superior to medical therapy alone for the treatment of hemodynamically significant (>70%) atherosclerotic renal artery stenosis, diagnosed by duplex doppler ultrasonography and confirmed by magnetic resonance angiography, in terms of avoidance of the progression of renal damage, control of hypertension and in reducing the cerebro and cardiovascular complications.

DETAILED DESCRIPTION:
Atherosclerotic renovascular disease (ARVD), due to renal hypoperfusion caused by mono or bilateral renal artery stenosis (RAS), is a increasing cause of chronic kidney disease and many elderly patients start dialysis due to ARDVD. Moreover ARVD is frequently progressive and reduces life-expectancy more than other causes of end stage renal disease, with a mortality rate higher than in patients with stable angina, similar to that of patients operated for colon cancer.

Unfortunately, there is not a definite therapy to cure this disease, despite important advancements in both medical therapy and in interventional radiology. Aim of the study is to see whether percutaneous transluminal interventional radiology plus stenting (PTRS) of the renal artery offers more, in terms of both preventing the progression of renal failure and controlling the hypertension, compared with the medical therapy addressed to control hypertension, improve the dyslipidemic profile and optimise the platelet anti-aggregant therapy, following the most recent guidelines. The eligible patients will be centrally randomized to:

1. medical treatment with hypotensive drugs (all class of hypotensive agents will be used according to single-center experience including drugs agent on renin-angiotensin-aldosterone-system, when permitted), lipid lowering therapy (namely all class of statins-or hydroxymethylglutaryl-coA reductase inhibitors)and anti-platelet (acetylsalicylate and/or ticlopidine or clopidrogel according to single-center experience) or to
2. the same medical therapy, as previously described in group a, associated with PTRS, according to a standardized protocol, with a follow up at 2 years extended to other 2 years

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 80 years
* Presence of ostial renal artery stenosis ≥ 70% (determined by Duplex Doppler ultrasonography and confirmed by Magnetic Resonance valuated by at least two experienced operators)
* Serum creatinine ≤ 3 mg/dl and/or creatinine clearance (Modification of Diet in Renal Disease, MDRD formula)≥ 30 ml/min, defined as stage 3 or greater CKD based on National Kidney Foundation classification
* Longitudinal ultrasonographic diameter of the stenotic kidney ≥ 8 cm
* Blood pressure values ≤ 150/90 mmHg with the use of less than four hypotensives drugs

Exclusion Criteria:

* Age > 80 years
* Other well-known nephropathy cause of renal failure
* Duplex doppler ultrasonography Resistive Index values >0.8
* Total occlusion of renal artery lumen
* Occurrence of cerebral or cardiac vascular diseases in the 6 months before the enrolment in the study
* Malignancy with a life expectation less than one year
* Previous documented cholesterol thrombo embolization episodes (clinically, bioptically or instrumentally)
* Liver failure
* Cardiac failure (NYHA IV class) or instable angina
* Well-known intolerance or contraindications to the use of iodinated contrast media, to statins or to anti platelets drugs
* Previous renal angioplasty
* Pregnancy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-10; Primary Completion 2008-09 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Death, Initiation of dialysis therapy or either serum creatinine increase more than 20% or reduction by > 20% in estimated clearance of creatinine (with MDRD formula) | 0.5, 1 and 2 years follow up plus extended 4 yrs

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure values at 0.5, 1 and 2 yrs follow up, with an extended follow up after 2 yrs | 0.5, 1 and 2 years follow up plus extended 4 yrs
Number of hypotensive drugs | 0.5, 1 and 2 years follow up plus extended 4 yrs
Results of renal scintigraphy | 0.5, 1 and 2 years follow up plus extended 4 yrs
Incidence of complications due to interventional manoeuvres | 0.5, 1 and 2 years follow up plus extended 4 yrs
Changes in the incidence of vascular complications in extra-renal districts | 0.5, 1 and 2 years follow up plus extended 4 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Scarpioni, Principal Investigator — Divisione Nefrologia e Dialisi, "Guglielmo da Saliceto" Hospital, Azienda USL Piacenza, Italy; Emanuele Michieletti, Principal Investigator — U.O. Radiologia II "Guglielmo da Saliceto" Hospital, Piacenza
Locations (1):
- Divisione di Nefrologia e Dialisi, "Guglielmo da Saliceto" Hospital, Azienda USL Piacenza, Piacenza, Piacenza, Italy

REFERENCES:
- [Result] Scarpioni R, Michieletti E, Cristinelli L, Ugolotti U, Scolari F, Venturelli C, Cancarini G, Pecchini P, Malberti F, Maroldi R, Rozzi G, Olivetti L. Atherosclerotic renovascular disease: medical therapy versus medical therapy plus renal artery stenting in preventing renal failure progression: the rationale and study design of a prospective, multicenter and randomized trial (NITER). J Nephrol. 2005 Jul-Aug;18(4):423-8. PMID 16245247